CLINICAL TRIAL: NCT01525212
Title: Double-Blinded, Placebo-controlled, Multiple Ascending Dose Study to Evaluate the Antiviral Activity, Safety, Tolerability, and Pharmacokinetics of BMS-929075 in Treatment Naive Subjects Infected With Hepatitis C Virus Genotype 1
Brief Title: Multiple Ascending Dose Study of BMS-929075 in Hepatitis C Virus (HCV) Infected Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI457-002
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: BMS-929075 (≤ 25 mg) OR Placebo matching BMS-929075 (Experimental)
  Interventions: Drug: BMS-929075; Drug: Placebo matching BMS-929075
- Arm 2: BMS-929075 (≤ 100 mg) OR Placebo matching BMS-929075 (Experimental)
  Interventions: Drug: BMS-929075; Drug: Placebo matching BMS-929075
- Arm 3: BMS-929075 (≤ 400 mg) OR Placebo matching BMS-929075 (Experimental)
  Interventions: Drug: BMS-929075; Drug: Placebo matching BMS-929075
- Arm 4: BMS-929075 (≤ 800 mg) OR Placebo matching BMS-929075 (Experimental)
  Interventions: Drug: BMS-929075; Drug: Placebo matching BMS-929075

INTERVENTIONS:
Drug: BMS-929075 — Oral Suspension, ≤ 25 mg, Once daily, 3 days
  Arms: Arm 1: BMS-929075 (≤ 25 mg) OR Placebo matching BMS-929075
Drug: BMS-929075 — Oral Suspension, ≤ 100 mg, Once daily, 3 days
  Arms: Arm 2: BMS-929075 (≤ 100 mg) OR Placebo matching BMS-929075
Drug: BMS-929075 — Oral Suspension, ≤ 400 mg, Once daily, 3 days
  Arms: Arm 3: BMS-929075 (≤ 400 mg) OR Placebo matching BMS-929075
Drug: BMS-929075 — Oral Suspension, (≤ 800 mg, Once daily) OR (≤ 400 mg, Twice daily), 3 days
  Arms: Arm 4: BMS-929075 (≤ 800 mg) OR Placebo matching BMS-929075
Drug: Placebo matching BMS-929075 — Oral Suspension, 0 mg, Once daily, 3 days
  Arms: Arm 1: BMS-929075 (≤ 25 mg) OR Placebo matching BMS-929075; Arm 2: BMS-929075 (≤ 100 mg) OR Placebo matching BMS-929075; Arm 3: BMS-929075 (≤ 400 mg) OR Placebo matching BMS-929075
Drug: Placebo matching BMS-929075 — Oral Suspension, 0 mg, (Once daily for ≤ 800 mg group) OR (Twice daily for ≤ 400 mg group), 3 days
  Arms: Arm 4: BMS-929075 (≤ 800 mg) OR Placebo matching BMS-929075

SUMMARY:
The purpose of this study is to determine the change from baseline in HCV Ribonucleic acid (RNA) on Day 4 following three days of dosing with BMS-929075 in chronically genotype subtype 1a and 1b HCV infected subjects

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 to 65 years, inclusive
* Subjects who are naive to HCV treatment, defined as no previous exposure to an Interferon (IFN), Ribavirin (RBV); or any HCV-specific direct acting antiviral or experimental therapy
* HCV genotype 1a or 1b only
* HCV RNA viral load of ≥ 100,000 IU/mL
* Have one of the following: i) Documented Fibrotest score of ≤ 0.72 and AST to platelet ratio index (APRI) ≤ 2; or ii) Documented liver biopsy within 12 months preceding Day 1 showing absence of cirrhosis
* Body Mass Index (BMI) of 18.0 to 35.0 kg/m2, inclusive

Exclusion Criteria:

* Any significant acute or chronic medical illness
* History of adrenal gland disease, including but not limited to adrenal insufficiency or Cushing's syndrome
* Current or recent (within 3 months of study drug administration) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* Any gastrointestinal surgery that could impact upon the absorption of study drug
* Positive for hepatitis B surface antigen (HBsAg)
* Positive for Human Immunodeficiency Virus (HIV) -1 and/or -2 antibodies
* Smoking > 10 cigarettes per day
* Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) > 5x upper limit of normal (ULN)
* Total Bilirubin ≥ 1.5x ULN
* Hemoglobin < 10 g/dL
* Platelets < 75,000 cell/μL
* ALC (absolute lymphocyte count) < 1000 cell/μL
* Creatinine clearance (as estimated by method of Cockcroft and Gault) less than 60 mL/min

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
HCV RNA level on Day 4 | Within 4 days after the first dose

SECONDARY OUTCOMES:
Maximum decrease from baseline in plasma HCV RNA levels during the period from Day 1 to Day 28 | Days 1-28
Time course of the change from baseline in plasma HCV RNA levels and the time of maximum decrease during the period of Day 1 through Day 28 | Days 1-28
Safety assessments will be based on medical review of adverse event reports and the results of vital sign measurements, ECGs, physical examinations, and clinical laboratory tests | Days 1-28 (with SAE from screening to Day 30)
Maximum observed plasma concentration (Cmax) of BMS-929075 derived from plasma concentration versus time | Day 1 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h), Day 2, and Day 3 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h,24h, 36h, 48h and 72h)
Minimum observed plasma concentration (Cmin) of BMS-929075 derived from plasma concentration versus time | Day 1 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h), Day 2, and Day 3 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h,24h, 36h, 48h and 72h)
Trough observed plasma concentration (Ctrough) of BMS-929075 derived from plasma concentration versus time | Day 1 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h), Day 2, and Day 3 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h,24h, 36h, 48h and 72h)
Time of maximum observed plasma concentration (Tmax) of BMS-929075 derived from plasma concentration versus time | Day 1 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h), Day 2, and Day 3 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h,24h, 36h, 48h and 72h)
Area under the concentration-time curve in one dosing interval [AUC(TAU)] of BMS-929075 derived from plasma concentration versus time | Day 1 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h), Day 2, and Day 3 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h,24h, 36h, 48h and 72h)
Plasma half-life (T-HALF) of BMS-929075 derived from plasma concentration versus time | Day 1 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h), Day 2, and Day 3 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h,24h, 36h, 48h and 72h)
Protein Binding (PB) of BMS-929075 derived from plasma concentration versus time | Day 3 (0h and 2h)
Fraction of free drug in plasma (fu) of BMS-929075 derived from plasma concentration versus time | Day 1 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h), Day 2, and Day 3 (0h, 0.5h, 1 h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h,24h, 36h, 48h and 72h)
The relationship between antiviral activity and measures of exposure to BMS-929075 | Days 1-6

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- Australia (3):
  - Local Institution, Herston, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Melbourne, Victoria

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx